## Design and Implementation of a Nutritional Intervention in Patients With Oropharyngeal Dysphagia

NCT02959450

October 10th, 2021

## Statistical analysis

The data are presented as mean ± standard deviation or median with interquartile range [25th- 75th percentile], depending of data distribution. The Shapiro-Wilk test for proper parametric or non-parametric test was performed. Differences between groups at baseline were evaluated with Student's t-test or U Mann-Whitney test for continuous variables and proportions were compared using the Chi2 or Fisher test. Two analyses were performed to evaluate the effect of the nutritional intervention: an intention-to-treat analysis (considering all of the participants) and per-protocol analysis (considering participants who finished the follow-up). Missing data were imputed with the multivariate imputation. For the intention- to-treat analysis, we imputed five complete data sets and pooled the results for the analysis. For postintervention comparison within-groups, a paired Student-t or Wilcoxon matchedpairs signed rank tests were performed. Also changes between baseline and final intervention in oral intake, body weight and HGS were obtained between groups and were compared with the Mann-Whitney U test, according to the nonparametric distribution of the data. A p-value <0.05 was considered statistically significant. The data were analyzed using the Statistical Package for the Social Sciences (SPSS®) version 25.